CLINICAL TRIAL: NCT01195181
Title: Improvement of the Surveillance and Control of Liver Disease and Complication Due to Chronic Hepatitis C: Project A) Antiviral Drugs Use, Efficacy, Safety and Costs; Project B) Kinetics of Virological Response.
Brief Title: Different PEG-interferon and Ribavirin Schedules for Chronic Hepatitis C in the Real Clinical Practice.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera di Padova (Other)
Collaborators: Regione Veneto (Other); University of Padova (Other)
Responsible Party: Liliana Chemello, M.D, Ph.D., Scientific Director, Department of Clinical and Experimental Medicine, University of Padua. Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEPCOVE protocol; DRG N.2920/2002 (Other Grant/Funding Number: Regione Veneto)
Record Dates: First submitted 2010-08-31; First posted 2010-09-06 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Hepatitis C Virus; Chronic Liver Disease; Viral Hepatitis; Therapeutic Uses; Antiviral Agents
Keywords: peginterferon alfa 2a and 2b type; ribavirin; chronic hepatitis C; antiviral therapy cost/efficacy; viral kinetics
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- peginterferon alfa-2a plus ribavirin (Active Comparator): patients will receive a fixed dose of 180ug/week of peginterferon alfa-2a plus ribavirin at 15mg/kg/daily.
  Interventions: Drug: peginterferon plus ribavirin
- peginterferon alfa-2b plus ribavirin (Active Comparator): patients will receive a weight adjusted dose (1,5ug/kg) from 50 to 150ug/week of peginterferon alfa-2b (standard dose) or a lower dose (1,0ug/kg) at physician discretion (randomization list available only for 100 cases) plus ribavirin at 15mg/kg/daily.
  Interventions: Drug: peginterferon plus ribavirin

INTERVENTIONS:
Drug: peginterferon plus ribavirin — peginterferon alfa-2a at 180ug/week (preempt syringe, sc) or peginterferon alfa-2b at 1,5 ug/kg/week (standard dose) or at 1,0 ug/kg/week (lower dose)(preempt pen, sc) for 24 or 48 week in relation to HCV genotype plus ribavirin (capsules, po) at 15mg/kg/daily combination therapy.
  Other Names: Pegasys; PegIntron; Copegus; Rebetol

SUMMARY:
Hepatitis C virus (HCV) infection provokes thousands of deaths every year all over the world, being the major cause of progressive liver disease, primary hepatic cancer and liver transplantation. Today, a "curative" therapy is available, that can eradicate the viral infection and determine the regression of liver fibrosis, also in cirrhotic subjects.

The current standard-of-care for HCV chronic infection is combination therapy with peginterferon (P-IFN) and ribavirin (RBV). However, this treatment is not only expensive but determines several side effects, that can reduce drug tolerance and hence, patient adherence to therapy. There are two types of available P-IFN on the market: P-IFN alfa-2a (Pegasys®, F.Hoffmann-La Roche) administered at a flat-dose of 180 mcg/week and P-IFN alfa-2b (PegIntron®, Schering-Plough) given at a weight-based dose of 50 to 150 mcg/week. Since only a single amino acid differentiates these types of IFN, administration strategies depend on their pegilation with molecules of 40 or 12kDa, respectively, that accounts for differences in the pharmacokinetic and pharmacodynamic drug-profile and influences probably also bioactivity. No comparative data are available on the benefits and costs of the licensed Peg-IFN plus RBV for the treatment of HCV infection in the real clinical practice, even if, the benefit and favourable cost-efficacy of this antiviral therapy is well established and of large consensus. Recently, the first randomized controlled mega-trial to compare antiviral therapeutic efficacy in naïve patients with HCV-genotype 1 infection during different regimens of P-IFN alfa-2b (at low and standard-dose) and P-IFN alfa-2a plus RBV, has been published, confirming a similar efficacy, of around 40%, obtained with the three schedules evaluated.

In Italy, a regional program on the Surveillance and Control of HCV Infection, set up by the Regional Health Councillorship, has led to the development of a clinical and epidemiological observatory, constituted by a network of liver tertiary centres (Hepatological Cooperative Network of Veneto, HepCoVe). This collaborative group is connected on-line by a common database that, since 2003, has prospectively collected data on a cohort of more than 3000 patients with chronic HCV infection and, among them, of 506 naïve subjects that consecutively underwent combination therapy with P-IFN alfa-2a or alfa-2b plus RBV.

The aim of this study was to rationalize and improve the social regional health program on antiviral treatment of chronic hepatitis C by assessing the different schedules utilization of P-IFN plus RBV as well as the respective therapeutic effectiveness, safety and costs in the real clinical practice (Project A).

DETAILED DESCRIPTION:
(Project B) To evaluate the viral kinetic decay during antiviral combination therapy with P-IFN alfa-2a and 2b type plus ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Naive adult subject
* active HCV infection (HCV-RNA positive)
* histological/biochemical signs of chronic hepatitis or compensated cirrhosis
* willingness of treatment

Exclusion Criteria:

* autoimmune disorders
* severe depression or psychiatric disease
* previous decompensation of cirrhosis
* gastroesophageal bleeding
* hepatocellular carcinoma
* major disease with a life expectancy of less than 5 years
* pregnancy or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of real dose drugs intake in relation to sustained virological response (SVR). | Measurement of HCV-RNA at 24° week after therapy withdrawal.
  Project A) The analysis will describe the efficacy (SVR) and costs of the 3 different antiviral schedules proposed.

SECONDARY OUTCOMES:
Description of the profile of the virus decay during antiviral therapy in relation to virological response. | Measurement of HCV-RNA during therapy in relation to negativity at 24° week after therapy withdrawal.
  Project B) The analysis will evaluate the kinetics of virological response obtained with the two peginterferons plus ribavirin by HCV-RNA quantification (Cobas,TaqMan, Roche) at basal time and at 1°,4°,12°,24°,36°,48° week during therapy and at 24° week after therapy withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: liliana chemello, M.D., Ph.D., Study Chair — University of Padova; luisa cavalletto, M.D., Ph.D., Principal Investigator — Azienda Ospedaliera di Padova
Locations (1):
- Department of Clinical and Experimental Medicine, Out-patients Hepatologic Unit, Azienda Ospedaliera di Padova., Padua, Italy

REFERENCES:
- [Background] Alberti A, Chemello L. and Benvegnù L. Natural history of hepatitis C. J Hepatol. 1999;31:17. Stroffolini T, Andreone P, Andriulli A et al. Characteristics of hepatocellular carcinoma in Italy. J Hepatol. 1998;29:944. Veldt BJ, Heathcote EJ, Wedemeyer H, et al. Sustained virological response and clinical outcomes in patients with chronic hepatitis C and advanced fibrosis. Ann Inter Med. 2007;147:677. Russo MW. and Fried MW. Side effects of therapy for chronic hepatitis C. Gastroenterology 2003;124:1711. Fried MW, Shiffman ML, Reddy KR, et al. Peginterferon alfa-2a plus ribavirin for chronic hepatitis C virus infection. N Engl J Med. 2002;347:975. Manns MP, McHutchison JG, Gordon SC, et al. Peginterferon-alfa-2b plus ribavirin compared with interferon alfa-2b plus ribavirin for initial treatment of chronic hepatitis C: a randomized trial. Lancet 2001; 358: 958. Caliceti P. Pharmacokinetics of pegylated interferons: What is misleading? Dig Liver Dis. 2004;36:S334. Di Bisceglie AM, Ghalib RH, Hamzeh FM. and Rustgi VK. Early virologic response after peginterferon alpha-2a plus ribavirin or peginterferon alpha-2b plus ribavirin treatment in patients with chronic hepatitis C. J Viral Hepatitis. 2007;14:721. Malone DC, Tran TT. and Poordad FF. Cost-efficacy analysis of peginterferon alfa-2b plus ribavirin compared with peginterferon alfa-2a plus ribavirin for the treatment of chronic hepatitis C. J Manag Care Pharm. 2005;11: 687. McHutchinson JG, Lawitz EJ, Shiffman ML, for the IDEAL Study Team. Peginterferon Alfa-2b or Alfa-2a with Ribavirin for treatment of hepatitis C infection. NEJM 2009;361(6):580. Hadziyannis SJ, Sette H.Jr, Morgan TR, et al. Peginterferon-alpha2a and ribavirin combination therapy in chronic hepatitis C: a randomized study of treatment duration and ribavirin dose. Ann Intern Med. 2004;2;140(5):346.